CLINICAL TRIAL: NCT01183559
Title: Induction Therapy for Locally Advanced, Resectable Cancer of the Esophagus, Gastroesophageal (GE) Junction and Gastric Cancer: A Phase I Trial of ZD6474 (Zactima, Vandetanib), Paclitaxel, Carboplatin, 5-Fluorouracil, and Radiation Therapy Followed by Surgery
Brief Title: A Trial of ZD6474, Paclitaxel, Carboplatin, 5-Fluorouracil, and Radiation Therapy Followed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCCC IRB 07-017; NCT00462033 (obsolete NCT alias)
Record Dates: First submitted 2010-08-13; First posted 2010-08-17 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Cancer of the Esophagus; Adenocarcinoma of the Gastroesophageal Junction; Cancer of the Stomach
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — vandetanib; Fluorouracil; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vandetanib (Other): Vandetanib 100 mg (6 patients) or 200 mg (3 patients) orally daily during the conventional 3D-guided conformal radiation therapy plus chemotherapy with carboplatin (AUC 5) on days 1 and 29, paclitaxel 50 mg/m2 i.v. weekly on days 1, 8, 15, 22, 29; and continuous infusion of 5-fluorouracil at 225 mg/m2 for 96 hours Monday-Friday during the radiation.
  Interventions: Drug: Vandetanib; Drug: 5 Fluorouracil (FU); Drug: Carboplatin; Drug: Paclitaxel; Radiation: External Beam Radiation Therapy (RT)

INTERVENTIONS:
Drug: Vandetanib — Vandetanib 100mg orally escalating to doses of 200 mg daily 7 days a week until completion of radiation therapy
  Other Names: ZD6474; Zactima
Drug: 5 Fluorouracil (FU) — 5-FU 225 mg/m2/day continuous infusion over96 hours during radiation therapy
  Other Names: 5-FU
Drug: Carboplatin — Carboplatin AUC=5 days 1 and 29 during radiation therapy
Drug: Paclitaxel — Paclitaxel 50 mg/m2 days 1, 8, 15, 22, 29 during radiation therapy
  Other Names: Taxol
Radiation: External Beam Radiation Therapy (RT) — External Beam Radiation Therapy(XRT)to a total dose of 4,500 centiGray (cGy) (180 cGy fractions daily) Monday through Friday for five weeks
  Other Names: XRT; RT

SUMMARY:
The purpose of the study is to determine the most tolerable and safe dose of ZD6474 (Zactima, Vandetanib) when given with standard chemotherapy, radiation therapy and surgery in patients with cancer of the esophagus

DETAILED DESCRIPTION:
Epidermal Growth Factor Receptor (EGFR) is known to be an important prognostic factor for patients with esophageal cancer-overexpression is associated with a worse prognosis. Review of the literature demonstrates presence of EGFR expression in up 90% of cases of esophageal cancer. Additionally, Vascular Endothelial Growth factor (VEGF) is commonly overexpressed in esophageal cancer (especially adenocarcinoma) and is linked to the transition from Barrett's esophagus to invasive adenocarcinoma. Esophageal cancers with overexpression of VEGF are associated with a worse prognosis and poorer response to conventional chemoradiation.

Therefore, we feel it would be valuable to add an inhibitor of EGFR and VEGFR to the therapy of esophageal cancer to increase the rate of pathologic complete response and thus improve overall survival. In current trials of ZD6474 in combination with chemotherapy, the dose has been 300mg. We will perform a phase I trial in which we will dose-escalate ZD6474 to determine if this drug is tolerable in combination with cytotoxic chemotherapy and external beam radiation therapy. This would be the first trial in humans in which f these three modalities would be combined. We will determine the maximum tolerated dose of ZD6474 in this small trial and then hope to perform a larger phase II trial, perhaps in the context of the Radiation Therapy Oncology Group (RTOG).

ELIGIBILITY:
Inclusion criteria:

* Histologically documented carcinoma of the esophagus, gastroesophageal junction, or stomach for which chemo/radiation therapy is appropriate.
* Potentially resectable esophageal, Gastroesophageal junction carcinoma, or stomach carcinoma
* Eastern Cooperative Oncology Group Performance Status = 0-2
* No evidence of distant metastases
* Age 18 or greater
* Signed informed consent
* Willingness to practice adequate contraception in women of childbearing potential (WOCBP). Contraception must be continued for one month following discontinuation of the study drugs. Females who are WOCBP must have negative pregnancy test within 7 days of the first treatment. WOCBP includes any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is postmenopausal (defined as amenorrhea >=12 consecutive months, or women on hormone replacement therapy (HRT) with documented plasma follicle-stimulating hormone (FSH) level >35 mIU/mL). Even women who are using oral, implanted, or injectable contraceptive hormones or mechanical products (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g. vasectomy), should be considered to be WOCBP. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion criteria:

* Previous radiation therapy to chest or upper abdomen.
* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol.
* Impaired cardiac function at baseline, including any of the following:
* Clinically significant cardiac event such as myocardial infarction; New York Heart Association (NYHA) classification of heart disease >2 within 3 months before registration; or presence of cardiac disease that, in the opinion of the Investigator, increases the risk of ventricular arrhythmia.
* Inadequate pulmonary and cardiac function to tolerate surgery (see section 12): left ventricular ejection fraction <45% and/or a positive stress test; or Forced Expiratory Volume (FEV1) of <1.1 liters.
* History of arrhythmia (multifocal premature ventricular contractions (PVCs), bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) which is symptomatic or requires treatment or asymptomatic sustained ventricular tachycardia. Atrial fibrillation, controlled on medication is not excluded.
* Previous history of QTc prolongation as a result from other medication that required discontinuation of that medication.
* Congenital long QT syndrome, or 1st degree relative with unexplained sudden death under 40 years of age.
* Presence of left bundle branch block (LBBB).
* QTc with Bazett's correction that is unmeasurable, or >or= 480 msec on screening ECG. If a patient has QTc >or= 480 msec on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart). The average QTc from the three screening ECGs must be <480 msec in order for the patient to be eligible for the study).
* Any concomitant medication that may cause QTc prolongation, induce Torsades de Pointes or induce CYP3A4 function
* Hypertension not controlled by medical therapy (systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 100 mm Hg)
* Women who are currently pregnant or breast feeding.
* Previous or current malignancies within the last 5 years, with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
* Receipt of any investigational agents within 30 days prior to commencing study treatment.
* Uncontrollable diarrhea that may affect the ability of the patient to absorb ZD 6474 or tolerate side-effects.

Laboratory results:

* Adequate bone marrow function as defined by granulocyte count < 1500/mm^3 and platelet count < 100,000
* Serum bilirubin >1.5x the upper limit of reference range (ULRR)
* Serum creatinine >1.5 x ULRR or creatinine clearance < 50 mL/minute (calculated by Cockcroft-Gault formula.)
* Potassium < 4.0 mmol/L despite supplementation; serum calcium (ionized or adjusted for albumin,) or magnesium out of normal range despite supplementation.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 2.5 X ULRR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-08-07 (Actual); Primary Completion 2010-11 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Igor Astsaturov,, M.D., Ph.D., Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Details: Patients were accrued between March 2009 and August 2010 at Fox Chase Cancer Center outpatient medical oncology clinics.
Pre-assignment Details: Resectable stage II-III esophageal and GE junction carcinomas;staging by CT and PET scans, endoscopic ultrasound. Patients with a history or presence of ventricular dysfunction, ventricular or atrial arrhythmias; heart block; congestive heart failure; recent myocardial infarction,unstable angina, or uncontrolled hypertension were excluded
Groups:
- Vandetanib: All patients were treated with vandetanib with dose escalation from 100 mg (dose level 1) to 200 mg (dose level 2) orally daily for the duration of radiation therapy
Period: Overall Study
Arm/Group | Vandetanib
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vandetanib
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years]
  Years | 58 [35 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Tumor site type [Number; unit: Participants] — Middle third, lower third, GE junction
  Participants
    Middle third | 1
    Lower third | 6
    GE junction | 2
Primary Site of Disease [Number; unit: Participants]
  Esophagus | 2
  Gastroesophageal junction | 7

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Vandetanib
Description: To determine the maximum tolerated dose (MTD) of Vandetanib given concurrently with chemotherapy and radiation therapy followed by surgery (esophagectomy)evaluated by the frequency, severity and duration of adverse events that occur during treatment and for four weeks following surgery as measured by serial blood tests, electrocardiograms and physical assessments
Time Frame: Within 4 weeks of initiation of chemo/radiation therapy
Measure: Number; unit: milligrams
Groups:
- Vandetanib: All patients were treated with Vandetanib 100 mg QD (6 patients) or 200 mg daily (3 patients) orally daily during the conventional 3D-guided conformal radiation therapy plus chemotherapy with carboplatin (AUC 5) on days 1 and 29, paclitaxel 50 mg/m2 i.v. weekly on days 1, 8, 15, 22, 29; and continuous infusion of 5-fluorouracil at 225 mg/m2 for 96 hours Monday-Friday during the radiation.
Arm/Group | Vandetanib
Number analyzed (Participants) | 9
milligrams | 100

2. Secondary Outcome: The Number of Participants With Adverse Events
Description: To determine the safety and tolerability of Vandetanib when given in combination with chemotherapy and radiation therapy as evaluated by serial blood tests, electrocardiograms, and physical assessments during therapy and for four weeks following surgery
Time Frame: Within 4 weeks of initiation of chemo/radiation therapy
Measure: Count of Participants; unit: Participants
Groups:
- Vandetanib: All patients were treated with Vandetanib 100 mg QD (6 patients) or 200 mg QD (3 patients) orally daily during the conventional 3D-guided conformal radiation therapy plus chemotherapy with carboplatin (AUC 5) on days 1 and 29, paclitaxel 50 mg/m2 i.v. weekly on days 1, 8, 15, 22, 29; and continuous infusion of 5-fluorouracil at 225 mg/m2 for 96 hours Monday-Friday during the radiation.
Arm/Group | Vandetanib
Number analyzed (Participants) | 9
Participants | 2

ADVERSE EVENTS:
Time Frame: From initiation of Vandetanib therapy through 6 months
Description: Adverse events evaluated for severity and relationship to therapy using a grading system in which Grade 3 = severe, Grade 4 = life-threatening or disabling and Grade 5 = death
Arm/Group | Vandetanib
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vandetanib (N=9)
Aortic-enteric fistula (Gastrointestinal disorders) | 1 (1) — Grade 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vandetanib (N=9)
Anorexia (Gastrointestinal disorders) | 1 (1) — Grade 3
ALT-SGPT (Investigations) | 1 (1) — Grade 3
AST-SGPT (Investigations) | 1 (1) — Grade 3
Leukocyte, total WBC (Investigations) | 2 (2) — Grade 3
Mood alteration, Depression (Psychiatric disorders) | 1 (1) — Grade 3
Neutrophills, ANC/AGC (Investigations) | 1 (1) — Grade 3
Pain, upper abdomen (Gastrointestinal disorders) | 1 (1)
Sodium, serum low (hyponatremia) (Investigations) | 1 (1) — Grade 3
Syncope (Nervous system disorders) | 1 (1) — Grade 3
Mucositis (Gastrointestinal disorders) | 1 (1) — Grade 3
Stomach-Bronchial fistula (Gastrointestinal disorders) | 1 (1) — Grade 4

LIMITATIONS AND CAVEATS:
Study closed due to reaching the stated endpoint of determination of the phase II recommended and tolerated dose of Vandetanib

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No